CLINICAL TRIAL: NCT05335408
Title: A Randomized Controlled Trial on the Visual Function After Bilateral Implantation of Two Novel Extended Depth-of-Focus Intraocular Lenses
Brief Title: Evaluation of Visual Function After Bilateral Implantation of EDOF IOLs
Acronym: Vario-NL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL79042.068.21
Record Dates: First submitted 2022-03-31; First posted 2022-04-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Cataract Bilateral; Lens, Intraocular; Lens Implantation, Intraocular; Pseudophakia; Visual Acuity
Keywords: Extended depth of Focus intraocular lenses; Intermermediate visual acuity
MeSH Terms: conditions — Cataract; Pseudophakia

STUDY DESIGN:
Intervention Model Description: The study design is a single-center, double masked, prospective randomized clinical study. The study will be conducted at the University Eye Clinic Maastricht of the Maastricht University Medical Centre+ (MUMC+) in the Netherlands.
  The study consists of two study groups: Vario-group (implantation with the Acunex® Vario IOL) and the Vivity-group (implantation with the Alcon AcrySof® IQ Vivity® IOL). A total of 32 patients will be randomized into either the Vario-group or the Vivity-group at a 1:1 ratio. Patients and study-optometrists will be masked. Surgeons are impossible to mask, due to the difference in (optical) design between both IOLs. Patients will receive standard cataract extractions by experienced surgeons.
Who Masked: Participant
Masking Description: Study optometrists (who will perform the examinations)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vario-group (Experimental): Patients in this group recieve the Acunex Vario IOL bilaterally during the cataract surgery.
  Interventions: Device: Acunex Vario intraocular lens
- Vivity-group (Active Comparator): Patients in this group recieve the Alcon Acrysof IQ Vivity IOL bilaterally during the cataract surgery.
  Interventions: Device: Alcon AcrySof IQ Vivity intraocular lens

INTERVENTIONS:
Device: Acunex Vario intraocular lens — This is an extended depth of focus IOL, made by Teleon Surgical B.V.
  Arms: Vario-group
Device: Alcon AcrySof IQ Vivity intraocular lens — This is an extended depth of focus IOL, made by Alcon.
  Arms: Vivity-group

SUMMARY:
Since intermediate vision is becoming increasingly important in our day-to-day tasks, a new IOL was introduced (Acunex Vario) with this objective in mind. This IOL provides excellent vision at far and intermediate distances up to 60 cm and with negligible photopic disturbances compared to conventional multifocal lenses. The Alcon AcrySof IQ Vivity IOL is designed to provide continuous vision from distance to intermediate while preserving contrast sensitivity and with a monofocal visual disturbance profile. So far, there are no published studies comparing these new IOL designs that offer an extended range of vision at far and intermediate distances.

Objective: The primary objective of this study is to compare the binocular uncorrected intermediate visual acuity (UIVA) at 66 cm under photopic conditions 3 months postoperatively, in a series of patients bilaterally implanted with the Vario IOL versus those bilaterally implanted with the Vivity IOL.

Study design: controlled double masked, randomized, prospective clinical trial Study population: patients of 18 years or older with bilateral cataracts that require cataract surgery.

Intervention: One group receives bilateral implantation with the Vario IOL and the other group receives bilateral implantation with the Vivity IOL.

Main study parameters: The main study parameter is the binocular UIVA at 66 cm under photopic conditions at 3 months postoperatively.

Hypothesis: The investigators hypothesise that bilateral implantation with the Vario IOL is non-inferior when compared to bilateral implantation with the Vivity IOL, with regards to binocular UIVA at 66 cm under photopic conditions 3 months postoperatively.

Cataract extraction in this study will proceed according to regular cataract surgery. As with any type of intraocular surgery, there is a possibility of complications due to anesthesia, drug reactions, and surgical problems. Postoperatively, there will be one extra postoperative visit, compared to standard cataract surgery follow-up. Spectacle-independency postoperatively, without photopic phenomena, is one of the major expected benefits when treating cataract (and presbyopia) with the implantation of the Vario or Vivity IOLs.

DETAILED DESCRIPTION:
INTRODUCTION AND RATIONALE

Nowadays, the most common types of intraocular lenses (IOLs) to correct aphakia after cataract surgery consist of monofocal, multifocal or extended depth of focus (EDOF) IOLs.

Current monofocal IOLs provide one focal point which will provide the patient with unaided vision at only one distance, which necessitate the need of glasses to correct vision at all other distances.

Multifocal IOLs (mIOLs) can be divided into bifocal-, trifocal- or quadrifocal IOLs, and provide patients with unaided vision at more than one distance, causing less spectacle-dependency after cataract surgery. Although mIOLs offer better unaided near vision and less spectacle dependency in comparison to monofocal IOLs, a well-known drawback of mIOLs is the occurrence of halos and glare and the inherent loss of contrast sensitivity because of their optical design. The potential decrease in quality of vision makes implantation of mIOLs less suitable in highly demanding patients or in cases of pre-existing pathology of the visual pathway (i.e., macular degeneration, optic neuropathy, post refractive surgery).

EDOF IOLs offer an extended range of focus and enable the patient to have a wider range of unaided vision in comparison to monofocal IOLs, especially from intermediate to far, while mIOLs have shown better near vision in comparison to EDOF IOLs.

Photic phenomena like halos and glare are regarded as the most important drawbacks of mIOLs and EDOF lenses. These photic phenomena can be explained due to the optical design where either diffractive or zonal refractive technology is applied. These photic phenomena become less apparent in a few months after neuroadaptation has taken place in the majority of cases. However, these phenomena can persist in some patients and are one of the main reasons for IOL explantation.

Since intermediate vision is becoming increasingly important in day-to-day tasks due to smartphone, tablet and laptop use, a new IOL was introduced with this objective in mind. The extended depth of focus IOL provides vision at far and intermediate distances up to 60 cm. Both the Acunex® Vario and the Alcon AcrySof® IQ Vivity® IOL consist of this EDOF optic design. The Acunex® Vario IOL design includes a sector-shaped near vision +1.5D addition located on the anterior surface of the IOL. The Alcon AcrySof® IQ Vivity® IOL consists of two anterior surface transition elements: the surface transition element, which includes a slightly elevated plateau for stretching the wavefront, and a small curvature change for shifting the wavefront. The last mentioned wavefront-shaping area stretches and shifts the wavefront resulting in an extended focal range of >1.5 D.

The Alcon AcrySof® IQ Vivity® IOL is a commonly used EDOF IOL and has been used for several years offering good visual outcomes in patients. Patients who received this IOL in the Maastricht University Medical Center+ (MUMC+) are satisfied with their vision quality and rarely complain about dysphotopsias after implantation. The Acunex® Vario IOL is a new EDOF IOL. According to prior preliminary results and pilot studies, this IOL demonstrates good results, including excellent distance and intermediate visual acuity, very low levels of dysphotopsia and high levels of postoperative patients satisfaction.

Both IOLs offer extended depth of focus and have similar results according to our own experience and prior research, but there are no published studies comparing these IOLs in a randomized controlled trial. The aim of this study is to compare the optical function, side effects and patient satisfaction after implantation of the Acunex® Vario and Alcon Acrysof® IQ Vivity® IOL in a controlled double masked, randomized, prospective clinical trial.

STUDY DESIGN

Patients will be examined pre-operatively and 1 week, and 1 and 3 months postoperatively. Besides a preoperative visit at which both eyes are examined, 4 postoperative visits are included when delayed sequential bilateral cataract surgery (DSBCS) is performed: week 1 visit for the first operated eye, week 1 visit for the second operated eye, and 1-, and 3-months visits at which both eyes will be examined in the same visit. In the event that immediately sequential bilateral cataract surgery (ISBCS) is performed the week 1 visit will be combined resulting in 3 postoperative visits. In both scenario's (ISBCS or DSBCS) both eyes are examined simultaneously at 1, and 3 months postoperatively in order to minimize the number of postoperative follow-up visits for patients. Consequently, with DSBCS, at 1 months postoperatively, the first eye will be 5 weeks after surgery and the second eye 3 weeks. At 3 months postoperatively, the first eye will be 13 weeks after surgery and the second eye 11 weeks. The investigators assume that this time difference does not affect the results. At the control visits, patients will receive a general ophthalmic examination, imaging of the eye and will be asked to fill-in patient questionnaires.

The duration of the study is 18 months, based on preparation of the study in the first 3 months, the inclusion of patients into the Randomized Controlled Trial (RCT) in the following 9 months, a follow-up of 3 months after IOL implantation and analysis of the data during the last 3 months of the study.

STATISTICAL ANALYSIS

All data will be collected in Castor, an electronic data capture (EDC) system designed for medical research, and exported to SPSS (IBM Corp., USA) and/or Excel (Microsoft, USA) software packages for data analysis. For the final analysis of the data, a per-protocol analysis is used. For the analysis, only patients who have completed the originally allocated treatment (i.e. bilateral implantation of the Alcon AcrySof® IQ Vivity® IOL or the Acunex® Vario IOL), will be included.

All qualitative variables will be summarized as the distribution of frequency, absolute and percentage. For all quantitative variables, descriptive statistics (including mean [or median], SD, minimum and maximum values) will be calculated for all necessary parameters. All data will be presented as means with standard deviation or proportions with percentages. The frequency and proportion of patients with postoperative medical and lens complications, and ocular/visual symptoms will also be reported. SPSS will be used to determine the differences between groups and between pre- and postoperative assessments and evaluate whether these are equal (within the non-inferiority margin of 0.1 logMAR). T-tests for independent samples will be used to evaluate to what extent the outcomes of both study-groups are comparable, considering a non-inferiority margin of 0.1 logMAR. Further, paired t-tests will be used to analyse the changes in visual acuities between the preoperative and postoperative visits.

The student's t-test requires normally distributed variables. If this assumption is not true, the more robust non parametric Wilcoxon rank sum test or Mann-Whitney U test, when appropriate, will be used. In all tests the threshold of statistical significance will be assumed equal to p=0.05

ELIGIBILITY:
Inclusion Criteria:

* Minimum 18 years of age
* Bilateral cataract
* Bilateral implantation of either Acunex® Vario IOL or the Alcon AcrySof® IQ Vivity® IOL
* Expected postoperative astigmatism ≤ 1.00 D (use of femtosecond laser assisted cataract surgery (FLACS) AK's tolerated up to 1.5 D of corneal astigmatism preoperative)
* Bilateral implantation of a non-toric Acunex® Vario IOL or a non-toric Alcon AcrySof® IQ Vivity® IOL
* IOL power calculation between +10.00 D and +30.0 D
* Expected postoperative best-corrected visual acuity of logMAR 0.3 or better
* Availability to undergo second eye surgery on the same day or else within 2 weeks of the first eye surgery
* Willing and able to comply with scheduled visits and other study procedures
* Signed informed consent

Exclusion Criteria:

* Previous corneal surgery and/or reshaping
* Corneal pathology (i.e., fuchs endothelial dystrophy (FED), irregular astigmatism, herpes simplex virus (HSV) keratitis
* Extensive age-related macular degeneration (atrophic or exudative age-related macular degeneration or numerous soft drusen) and post-intravitreal injection (IVI)
* Extensive visual field loss (eg. glaucoma, cerebral vascular accident (CVA), hemianopsia, etc.)
* Extensive diabetic retinopathy
* Amblyopia, strabismus, diplopia
* Pseudo exfoliation syndrome or other capsule or zonular abnormalities that could affect postoperative centration or tilt of the IOL
* Pupil abnormalities (non-reactive, tonic pupils, abnormally shaped pupils, or pupils that do not dilate at least 3.5 mm under mesopic /scotopic conditions)
* Cognitive cerebral or concentration disorders (e.g., dementia, Parkinson, stroke, etc.)
* Suturing of incision required at time of surgery
* Complications during surgery of the first eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2023-06-09 (Actual)

PRIMARY OUTCOMES:
Binocular uncorrected intermediate visual acuity | 3 months postoperatively
  The visual acuity will be measured at 66cm under photopic conditions

SECONDARY OUTCOMES:
Mono- and binocular uncorrected and corrected distance visual acuity | At week 1, 1 month and 3 months postoperatively
  The visual acuities will be measured at 4 meters under photopic conditions
Mean binocular distance-corrected intermediate visual acuity | At 1 and 3 months postoperatively
  The visual acuity will be measured at 66cm under photopic conditions
Mean binocular uncorrected near visual acuity and distaqnce corrected near visual acuity | At 1 and 3 months postoperatively
  The visual acuity will be measured at 40cm under photopic conditions
Binocular defocus curves | At 3 months postoperatively
  Under photopic conditions
Mean binocular constrast sensitivity | At 3 months postoperatively
  Under photopic and mesopic conditions
Complication profile including halos and glare | Up to 3 months postoperatively
  According to the 4-point likert scale (ranging from 'no' to 'very disturbing')
Questionnaires on patient satisfaction rate | Preoperatively and at 3 months postoperatively
  Using questionnaire: Catquest-NL, including different questions and answer options of satisfaction rate (4-point scale ranging from 'very dissatisfied' to 'very satisfied')
Questionnaires on patient difficulty rate | Preoperatively and at 3 months postoperatively
  Using questionnaire: Catquest-NL, including different questions and answer options of difficulties (4-point scale ranging from 'Very big difficulties' to 'no difficulties').
Questionnaires on occurence of optical complaints | At 3 months postoperatively
  Using questionnaires: QoV-NL, including different questions and answer options about how often the complaints happen (4-point scale ranging from 'never' to 'very often').
Questionnaires on the bothersome of optical complaints | At 3 months postoperatively
  Using questionnaires: QoV-NL, including different questions and answer options about how bothersome it is for the patient (4-point scale ranging from 'Not at all' to 'Very').
Questionnaires on spectacle independence | At 3 months postoperatively
  Using questionnaires: IOLSAT, including different questions and 5-point scale answer options ranging from 0 (Never) to 4 (Always)
Tilt and decentration intraocular lens | At 1 month postoperatively
  Using Optical Coherence Tomography scans

CONTACTS AND LOCATIONS:
Overall Officials: Rudy Nuijts, MD, PhD, Principal Investigator — University Eye Clinic Maastricht UMC+
Locations (1):
- Maastricht UMC+, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No
Only the results of the study will be published in report form and submitted for publication in appropriate journals in the international literature. IPD data will not be shared.

REFERENCES:
- [Background] Breyer DRH, Kaymak H, Ax T, Kretz FTA, Auffarth GU, Hagen PR. Multifocal Intraocular Lenses and Extended Depth of Focus Intraocular Lenses. Asia Pac J Ophthalmol (Phila). 2017 Jul-Aug;6(4):339-349. doi: 10.22608/APO.2017186. PMID 28780781
- [Background] Jonker SM, Bauer NJ, Makhotkina NY, Berendschot TT, van den Biggelaar FJ, Nuijts RM. Comparison of a trifocal intraocular lens with a +3.0 D bifocal IOL: results of a prospective randomized clinical trial. J Cataract Refract Surg. 2015 Aug;41(8):1631-40. doi: 10.1016/j.jcrs.2015.08.011. PMID 26432120
- [Background] de Vries NE, Nuijts RM. Multifocal intraocular lenses in cataract surgery: literature review of benefits and side effects. J Cataract Refract Surg. 2013 Feb;39(2):268-78. doi: 10.1016/j.jcrs.2012.12.002. PMID 23332253
- [Background] Vrijman V, van der Linden JW, van der Meulen IJE, Mourits MP, Lapid-Gortzak R. Multifocal intraocular lens implantation after previous corneal refractive laser surgery for myopia. J Cataract Refract Surg. 2017 Jul;43(7):909-914. doi: 10.1016/j.jcrs.2017.06.028. PMID 28823437
- [Background] Liu J, Dong Y, Wang Y. Efficacy and safety of extended depth of focus intraocular lenses in cataract surgery: a systematic review and meta-analysis. BMC Ophthalmol. 2019 Sep 2;19(1):198. doi: 10.1186/s12886-019-1204-0. PMID 31477053
- [Background] Kohnen T, Suryakumar R. Extended depth-of-focus technology in intraocular lenses. J Cataract Refract Surg. 2020 Feb;46(2):298-304. doi: 10.1097/j.jcrs.0000000000000109. PMID 32126045
- [Background] Webers VSC, Bauer NJC, Saelens IEY, Creten OJM, Berendschot TTJM, van den Biggelaar FJHM, Nuijts RMMA. Comparison of the intermediate distance of a trifocal IOL with an extended depth-of-focus IOL: results of a prospective randomized trial. J Cataract Refract Surg. 2020 Feb;46(2):193-203. doi: 10.1097/j.jcrs.0000000000000012. PMID 32126031
- [Background] Alio JL, Plaza-Puche AB, Fernandez-Buenaga R, Pikkel J, Maldonado M. Multifocal intraocular lenses: An overview. Surv Ophthalmol. 2017 Sep-Oct;62(5):611-634. doi: 10.1016/j.survophthal.2017.03.005. Epub 2017 Mar 31. PMID 28366683
- [Background] Erie JC, Simpson MJ, Bandhauer MH. A modified intraocular lens design to reduce negative dysphotopsia. J Cataract Refract Surg. 2019 Jul;45(7):1013-1019. doi: 10.1016/j.jcrs.2019.01.019. Epub 2019 Apr 16. PMID 31003799
- [Background] Ferreira TB, Ribeiro FJ. Prospective Comparison of Clinical Performance and Subjective Outcomes Between Two Diffractive Trifocal Intraocular Lenses in Bilateral Cataract Surgery. J Refract Surg. 2019 Jul 1;35(7):418-425. doi: 10.3928/1081597X-20190528-02. PMID 31298721